CLINICAL TRIAL: NCT02863172
Title: Molecular Basis for Variations in Hereditary Colorectal Cancer Syndromes
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA11-0567; 2015-00051016-Y1 (Other Grant/Funding Number: MD Anderson); 2016-00051406 (Other Grant/Funding Number: Eduardo Vilar-Sanchez, MD, PhD, Germline Precision Prevention in Adolescents)
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Hereditary Colorectal Cancer Syndrome
Keywords: Hereditary colorectal cancer syndrome; Questionnaires; Surveys; Blood sample; Saliva sample
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (about 2-3 tablespoons) drawn.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Consenting Proband Group: Questionnaires completed at baseline. Blood sample taken at baseline. Follow-up questionnaire completed at least 1 time in 5 years.
  Interventions: Behavioral: Questionnaires; Procedure: Blood Draw/Saliva Sample
- Family Members (MDA Registered Patients) Group: Health questionnaire completed at baseline. Blood sample taken at baseline. Follow-up questionnaire completed at least 1 time in 5 years.
  Interventions: Behavioral: Questionnaires; Procedure: Blood Draw/Saliva Sample
- Family Members (Not MDA Registered Patients) Group: Health questionnaire completed at baseline. Blood sample taken at baseline. Follow-up questionnaire completed at least 1 time in 5 years.
  Interventions: Behavioral: Questionnaires; Procedure: Blood Draw/Saliva Sample

INTERVENTIONS:
Behavioral: Questionnaires — Consenting Proband Group: Participants fill out questionnaires about work, family history, medical history, and health habits at baseline. It should take about 20 minutes to complete the questionnaires. Participants also complete a health and lifestyle questionnaire, which contains 20 questions for men and 22 questions for women. Questionnaire should take about 10 minutes to complete. Follow-up questionnaire at least 1 time in 5 years to update medical, cancer, and family history.
  Family Members (MDA Registered Patients) Group and Family Members (Not MDA Registered Patients) Group: Participants complete a health questionnaire, which collects information about their personal medical history, demographics (age, race, sex, and so on), and questions about their alcohol and tobacco use at baseline. Questionnaire should take about 20 minutes to complete. Participants complete follow-up questionnaire at least 1 time in 5 years to update their medical, cancer, and family history.
  Other Names: Surveys
Procedure: Blood Draw/Saliva Sample — About 2-3 tablespoons blood drawn. Participants may give a saliva sample instead.

SUMMARY:
Objectives:

1. To examine the variations in clinical features, survival outcomes, family history, and health behavior among proband patients who are known or suspected to have a hereditary colorectal cancer syndrome
2. To compare the clinical features, survival outcomes, and health behavior of the proband vs. his/her family members who may or may not be affected by the hereditary colorectal cancer syndrome
3. To explore for correlations between germline genetic variations in both the probands and family members with observed variations in the overall disease phenotype across probands and kindreds, within a given syndrome. Disease phenotype is defined to include: (1) clinicopathologic features including patient demographics and oncologic outcomes; (2) clinical manifestations of disease including the timing, spectrum and severity of CRC and extracolonic cancers. Genetic variations may include the specific codon mutated, the type of mutation and sequence alteration (e.g. nonsense, missense etc), chromosomal/gene copy number changes, and gene polymorphisms.
4. To explore for correlations between germline genetic variations in both the probands and family members with observed variations in somatic CRC tumor biology, including tumor pathology and other tumor molecular markers

DETAILED DESCRIPTION:
Participants:

Questionnaires:

If participant agrees to take part in this study, participant will fill out a some questionnaires about participant's work, family history, medical history, and health habits. If participant has already answered these questionnaires when participant was registered as a patient at MD Anderson, the study staff will give participant a copy and review participant's answers with participant for any updates or if participant has any questions. It should take about 20 minutes to complete the questionnaires.

Participant will also complete a health and lifestyle questionnaire, which contains 20 questions for men and 22 questions for women. This questionnaire should take about 10 minutes to complete.

Participant may be given the questionnaires electronically on REDcap (a secure, web-based application used to collect data for research studies that participant can access from participant's phone, tablet, or computer), over the phone (either with a member of the study staff asking questions or by using an electronic response system called IVR), at home through the mail, or in person by a member of the research staff at participant's MD Anderson visit. If mailed, a postage-paid return envelope will be provided for the return of the questionnaire.

Blood or Saliva Sample:

Blood (about 2-3 tablespoons) will be drawn. If possible, the blood will be drawn during an already scheduled blood draw to avoid additional needle sticks.

If participant is unwilling or unable to give a blood sample, participant may give a saliva sample instead. If participant is at MD Anderson, a saliva kit will be given to participant. If participant is not at MD Anderson, the kit will be mailed to participant with instructions for collecting the saliva sample and a prepaid envelope will be included to return the sample to the study staff.

The blood or saliva sample will be sent to the research laboratory of the study chairs at MD Anderson for testing.

Residual Tissue Collection:

If participant has tissue from procedures performed at MD Anderson, this tissue may be requested from participant's previous procedures for testing. If participant has had procedures done at another institution, participant may be asked to sign a waiver to allow the tissue from the outside institution to be sent to MD Anderson for testing.

Follow-Up Questionnaires:

Participant will also fill out a follow-up questionnaire at least 1 time in 5 years to update participant's medical, cancer, and family history. Each questionnaire will take approximately 20 minutes to complete.

Withdrawing from the Study:

Participant may withdraw from participation in this study at any time. If participant decides participant wants to stop taking part in this study, data collected about participant and data taken from the blood or saliva samples participant has provided up to the time participant withdraws will remain in study database and will be used for the purposes of the study.

Length of Study:

Participant's active participation on this study will be over after the blood, tissue, and/or saliva samples have been collected and participant has completed all of the questionnaires.

This is an investigational study.

Up to 2,000 patients and/or family members will take part in this study. All will be enrolled at MD Anderson.

Family Members:

Questionnaire:

Participant will complete a health questionnaire, which will collect information about participant's personal medical history, demographics (age, race, sex, and so on), and questions about participant's alcohol and tobacco use. This questionnaire should take about 20 minutes to complete.

Participant may be given the questionnaires electronically on REDcap (a secure, web-based application used to collect data for research studies that participant can access from participant's phone, tablet, or computer), over the phone (either with a member of the study staff asking questions or by using an electronic response system called IVR), at home through the mail, or in person by a member of the research staff at participant's family member's MD Anderson visit.

If mailed, a postage-paid return envelope will be provided for the return of the questionnaire.

Blood or Saliva Sample:

If participant agrees to take part in this study and participant is able to come to MD Anderson, blood (about 2-3 tablespoons) will be drawn.

If participant is unwilling or unable to give a blood sample, participant may give a saliva sample instead. If participant is at MD Anderson, a saliva kit will be given to participant. If participant is not at MD Anderson, the kit will be mailed to participant with instructions for collecting the saliva sample and a prepaid envelope will be included to return the sample to the study staff.

The blood or saliva sample will be sent to the research laboratory of the study chairs at MD Anderson for testing.

Outside Tissue Collection:

If participant has had a procedure done at a hospital, surgical center, or doctor's office outside of MD Anderson, participant may optionally be asked to sign a waiver to allow tissue stored at the outside hospital, surgical center, or doctor's office to be sent to researchers at MD Anderson.

Follow-Up Questionnaires:

Participant will also fill out a follow-up questionnaire at least 1 time in 5 years to update participant's medical, cancer, and family history. Each questionnaire will take approximately 20 minutes to complete.

Withdrawing from the Study:

Participant may withdraw from participation in this study at any time. If participant decides participant wants to stop taking part in this study, data collected about participant and data taken from the blood or saliva samples participant has provided up to the time participant withdraws will remain in study database and will be used for the purposes of the study.

Length of Study Participant's active participation on this study will be over after the blood, outside tissue and/or saliva samples have been collected and participant has completed all of the questionnaires.

This is an investigational study. Up to 2,000 patients and/or family members will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

Probands who meet the following criteria will be eligible:

1. Patient must have or is suspected to have a hereditary CRC syndrome
2. Patient must be at least 18 years of age at the time of study registration.
3. Patient must have sufficient command of the English language and mental capacity to provide consent

Family members who meet the following criteria will be eligible:

1. First- or second-degree relative of a registered MDACC patient who has met eligibility criteria for a Proband as defined above.
2. Family member must be at least 18 years of age at the time of study registration.
3. Family member must have sufficient command of the English language and mental capacity to provide consent

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants that have, or are suspected to have, a hereditary colorectal cancer syndrome registered at MD Anderson and family members.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-05-22 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Variations in Clinical Features Compared Between Proband Group and Family Member Group | 5 years
  Comparison made using 1-way ANOVA or Chi-squared tests.

SECONDARY OUTCOMES:
Variations in the Overall Disease Phenotype Between Proband Group and Family Member Group | 5 years
  Disease phenotype defined to include: (1) clinicopathologic features including patient demographics and oncologic outcomes; (2) clinical manifestations of disease including the timing, spectrum and severity of CRC and extracolonic cancers.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Qian N. You, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org